CLINICAL TRIAL: NCT04820075
Title: Efficacy of an Intervention to Improve the Preoperative Shower in Scheduled Surgery
Acronym: PRODOUCH'OP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: impossible to continue the study
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/0413/OB
Record Dates: First submitted 2021-03-12; First posted 2021-03-29 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-09

CONDITIONS: Surgery; Surgical Site Infection
Keywords: surgery; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: stepped wedged randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Process about performance of the preoperative shower (Other): Implementation of a process aimed at improving the preoperative shower in programmed surgery
  Interventions: Behavioral: improvement of preoperative shower

INTERVENTIONS:
Behavioral: improvement of preoperative shower — Process about preoperative shower

SUMMARY:
The aim of the project is to evaluate the effectiveness, on the skin cleanliness of the patient on arrival at the operating room, of an intervention aimed at improving the performance of the preoperative shower, for patients undergoing a planned surgical intervention in an orthopedic surgery department, digestive, gynecological, thoracic, or vascular.

DETAILED DESCRIPTION:
The project will be realized in 2 phases.

- The first phase of the project will consist of a sociological survey conducted with caregivers and patients in the care sectors participating in the study. This component sociological research will be carried out on the basis of in-depth interviews with caregivers (nurses and nursing assistants) from the departments concerned by research and patients. The expected sample, subject to data saturation, is 40 caregivers and 20 patients. These in-depth and non-directive interviews will be carried out by a sociologist and will aim to explore the way in which healthcare professionals see their activity professional, the relationship they maintain with the various members of the healthcare team, their perceptions of the body, privacy and hygiene of patients, but also to explore the representations of caregivers of the preoperative shower and of the relationship with caregivers during phases of explanation, possible help with the shower, and control of cleanliness cutaneous. These interviews will identify the representations of caregivers and patients with the aim of establishing a procedure for caregivers to improve care of the preoperative shower. In view of the statements of patients and caregivers concerning preparing for the preoperative shower and checking skin cleanliness during the Survey exploratory, it appears necessary to improve and formalize the protocol. Investigation will thus establish a base of knowledge necessary to establish a care procedure giving an account of the roles of each person, caregivers and patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 and over, and
2. scheduled for surgery (outpatient or full hospitalization) in one of the following specialties: orthopedics, digestive (including bariatric surgery), gynecological, thoracic, vascular, and
3. having read and understood the briefing note and not showing up for research.

Exclusion Criteria:

1. operated on urgently, or
2. operated on for an intervention other than orthopedics, gynecology, digestive surgery, vascular surgery, or
3. having received a toilet in bed, or
4. having expressed their opposition to the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
skin cleanliness | at the time of surgery
  The criterion for evaluating the effectiveness of the preoperative shower, consistent with national recommendations, is skin cleanliness, defined as the absence of macroscopic stains on the skin.

SECONDARY OUTCOMES:
occurrence of a surgical site infection | 30 days after surgery
  Occurrence of a surgical site infection (SSI)
postponement of surgery | Within 8 hours after shower
  Postponement of surgery due to insufficient cleanliness (no go)
need for detersion in the operating room | Within 8 hours after shower
  Need for debridement in the operating room for areas of surgery for which it is not systematic
patient's satisfaction regarding the preoperative shower | Within 1 month after shower
  Patient satisfaction with the preoperative shower
healthcare workers' satisfaction regarding the preoperative shower | Within 1 month after shower
  Satisfaction of caregivers responsible for the care of preoperative patients in the care unit and in the operating room
frequency of skin cleanliness assesment by healthcare workers | Within 8 hours after shower
  Verification of cleanliness by the caregiver (patient declarative data).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de ROUEN, Rouen, France

IPD SHARING:
Plan to Share IPD: No